CLINICAL TRIAL: NCT01097590
Title: A Randomized Placebo Controlled, Single Centre Study to Evaluate a Novel Leukapheresis Treatment in Patients With Ulcerative Colitis.
Brief Title: A Study to Evaluate a Leukapheresis Treatment in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IBD Column Therapies International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLA001; 461:2009/501 (Other: Medical Products Agency)
Record Dates: First submitted 2010-03-25; First posted 2010-04-01 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2010-03

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; leukapheresis treatment
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TLA Gut™ column (Experimental): The active column contain an engineered protein with the ability to specifically bind the inflammatory cells.
  Interventions: Device: Active TLA Gut™ column
- Placebo TLA Gut™column (Placebo Comparator): The placebo column is identical to the active column except it does not contain the engineered protein that specifically bind the inflammatory cells.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Active TLA Gut™ column — Five consecutive treatment sessions. The therapy will be administrated every second day.
  Other Names: TLA Gut™
  Arms: Active TLA Gut™ column
Device: Placebo — Five consecutive treatment sessions. The placebo therapy will be administrated every second day.
  Arms: Placebo TLA Gut™column

SUMMARY:
The purpose of this study is to determine whether a treatment of a novel leukapheresis column is safe and effective in patients with moderate to severe ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic and relapsing disease and is characterized by superficial inflammation in the colonic epithelium. The inflammation is maintained by continuous supply of inflammatory cells from the circulating blood to the intestinal mucosa.

Existing therapy e.g. corticosteroids and immunosuppressants are inadequate with an overall long-term remission rate of only 50-60%. Those treatments are also associated with severe side effects why there is a need of new therapies.

The aim of this study is to investigate a novel leukapheresis treatment with the potential to reduce the number of inflammatory cells homing to the gut mucosa. By drawing blood from the patient and pass it through the investigational column the inflammatory cells are removed. The blood, depleted of the inflammatory cells, is returned to the patient.

The treatment thus enable down-regulation of the inflammation and consequently the inflammation can heal. The treatment is called Tailored leukapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of active, moderate-to-severe, Ulcerative Colitis.

Exclusion criteria;

* Local intestinal treatments with suppositories, enemas or clysmas during the last 4 weeks
* Current daily smoking habits
* Other severe diseases as detailed in the protocol
* History of hypersensitivity to heparin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Expression level of MHC class II on antigen presenting cells. | change from baseline at day 5, 12, 28, 42 and 98.
  The primary outcome will be assessed by flow cytometry.

SECONDARY OUTCOMES:
The number of cells and/or expression level of gut homing and activation markers on lymphocytes and monocytes. Safety and tolerability. Clinical effect on signs and symptoms of the disease. | change from baseline at day 5, 12,28, 42, 98.
  The immunological analysis will be peformed by flow cytometry.
  The safety will be measured by recording adverese events at each visit.
  The disease activity will be assessed by using the Mayo Score Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eberhardson, Dr, Principal Investigator — Karolinska Universitetssjukhuset 171 76 Stockholm
Locations (1):
- Södersjukhuset, Stockholm, Sweden